CLINICAL TRIAL: NCT01290523
Title: Safety Profile Assessment of TheraSphere® Yttrium-90 Glass Microspheres Used for Treatment of Hepatocellular Carcinoma: A Pilot Study
Brief Title: Yttrium-90 Radioembolization With Glass Microspheres (TheraSphere) for Patients With Hepatocellular Carcinoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Off study clinical use of Y90 glass microspheres (TheraSphere)
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCSF-SIRT-HCC
Record Dates: First submitted 2011-02-01; First posted 2011-02-07 (Estimated); Results first posted 2015-08-25 (Estimated); Last update posted 2019-05-13 (Actual); Status verified 2019-04

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Yttrium-90 liver radioembolization (Experimental): Patients who receive liver-directed therapy with Yttrium-90 glass microspheres (TheraSphere)
  Interventions: Device: Selective internal radiation therapy of the liver with Yttrium-90 glass microspheres (TheraSphere)

INTERVENTIONS:
Device: Selective internal radiation therapy of the liver with Yttrium-90 glass microspheres (TheraSphere) — Administration of Yttrium-90 TheraSphere glass microspheres into the hepatic artery

SUMMARY:
This is a prospective pilot study that will document the clinical experience of 30 patients with unresectable hepatocellular carcinoma undergoing liver-directed therapy with Yttrium-90 glass microspheres (TheraSphere®).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hepatocellular carcinoma with liver-dominant disease. Diagnosis may be made by histo- or cyto-pathology, or by clinical and imaging criteria.
* The cancer is unresectable.
* All patients must be off all chemotherapeutic regimens for 30 days prior to and 30 days after TheraSphere treatment.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Age 18 years or older.
* Able to understand informed consent.

Exclusion Criteria:

* Evidence of potential delivery of greater than 16.5 mCi (30 Gy absorbed dose) of radiation to the lungs on either:

  * single TheraSphere administration; or
  * cumulative delivery of radiation to the lungs greater than 50 Gy over multiple treatments.
* Evidence of any detectable Tc-99m macroaggregated albumin flow to the stomach or duodenum, after application of established angiographic techniques to stop such flow.
* Previous radiation therapy to the lungs and/or to the upper abdomen
* Pregnancy
* Symptomatic lung disease.
* Significant extrahepatic disease representing an imminent life-threatening outcome.
* Active uncontrolled infection
* Any pre-treatment laboratory findings within 30 days of treatment demonstrating:

  * Aspartate or alanine aminotransferase level greater than 5 times upper normal limit.
  * Serum bilirubin greater than 2 mg/dl
  * Infiltrative tumor on imaging
  * Tumor volume greater than 70% of liver volume
  * Tumor volume greater than 50% of liver volume and serum albumin level less than 3 mg/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Fidelman, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Yttrium-90 radioembolization there were 14 total patients who signed consent and participated in the study. Enrollment started in May2010 and ended in June 2013.
Pre-assignment Details: A 2nd radioembolization treatment was allowed if patients had bilobar tumors and were willing to get repeated treatments.
Groups:
- Yttrium-90 Liver Radioembolization 1 Treatment: Patients who received 1 liver-directed therapy with Yttrium-90 glass microspheres (TheraSphere)
  Selective internal radiation therapy of the liver with Yttrium-90 glass microspheres (TheraSphere): Administration of Yttrium-90 TheraSphere glass microspheres into the hepatic artery
Period: Overall Study
Arm/Group | Yttrium-90 Liver Radioembolization 1 Treatment
Started | 14
Completed | 11
Not Completed | 3
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Arm/Group | Yttrium-90 Liver Radioembolization
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] — Age at time of first treatment
  years | 66 [58 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Adverse events of treatment with TheraSphere Yttrium-90 glass microspheres will be assessed within 6 months of treatment administration. Anticipated adverse events may include liver dysfunction, gastrointestinal ulcer formation, cholecystitis, pneumonitis, fatigue, nausea/vomiting, abdominal pain
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Yttrium-90 Liver Radioembolization
Number analyzed (Participants) | 14
participants | 3

2. Secondary Outcome: Radiographic Response by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) as assessed by MRI or CT:
  up to 5 lesions at baseline and sum longest diameters (SLD).
  * Complete Response (CR), -Target Lesions: Disappearance of all target lesions.
    -Non-target Lesions: disappearance of all non-target lesions and normalization of tumor marker level.
  * Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions;
  * Stable Disease (SD) < %30 decrease in the sum of the longest diameter of target lesions.
  * Progressive Disease (PD) -Target Lesions: > 20% increase in the SLD taking as reference the smallest SLD recorded since the treatment started (nadir) and minimum 5 mm increase over the nadir
  non-target lesions: Overall level of substantial worsening in non-target disease such that, even in presence of SD or PR in target disease, the overall tumor burden has increased sufficiently to merit discontinuation of therapy
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Yttrium-90 Liver Radioembolization
Number analyzed (Participants) | 14
Participants
  Complete Response (CR) | 0
  Partial Response (CR) | 5
  Stable Disease (SD) | 8
  Progressive Disease (PD) | 1

ADVERSE EVENTS:
Arm/Group | Yttrium-90 Liver Radioembolization
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 3/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Yttrium-90 Liver Radioembolization (N=14)
Fatigue (Injury, poisoning and procedural complications) | 3 (3) — NCI CTCAE grade 2 fatigue in two participants NCI CTCAE grade 1 fatigue in one participant

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No